CLINICAL TRIAL: NCT06257108
Title: Clinical Performance of Bulk-Fill Composite Using With Adhesives With or Without Chlorhexidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 01.04.2015/76
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-02

CONDITIONS: Class II Dental Caries
Keywords: Dentin bonding agents; chlorhexidine; antibacterial bonding; bulk-fill composite

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restorative group (Experimental): Class II restorations using chlorhexidine-containing bonding agent in Primary molars in children aged between 5-9 years.
  Interventions: Other: Class II Cavity Restorations
- Control Group (Active Comparator): Class II restorations using standard bonding agent in Primary molars in children aged between 5-9 years.
  Interventions: Other: Class II Cavity Restorations

INTERVENTIONS:
Other: Class II Cavity Restorations — The study involved a split-mouth design in which Ultradent PQ1 Bond (standard bond) and Ultradent Peak Universal Bond (chlorhexidine-containing bond) were used as the bonding agents, and Tetric N Ceram Bulk Fill composite was used as the restorative material for the restoration of primary molars with class II cavity.

SUMMARY:
This study aims to evaluate the clinical success of chlorhexidine-containing dentin bonding agent in primary molars with a 12-month follow-up. The research question is:

Is there a difference between the clinical evaluation results of deciduous teeth restored with dentin bonding agents containing and not containing chlorhexidine?

A total of 40 patients aged 5-9 years with at least two dentin caries in primary molars were included in the study. The study involved a split-mouth design in which the standard bond and chlorhexidine-containing bond as the adhesive agents. Bulk Fill composite was used as the restorative material for the restoration of primary molars with class II cavity. The evaluation of clinical success was performed by a calibrated observer according to the FDI criteria at months 3, 6, 9, and 12 after restoration.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical success of chlorhexidine-containing dentin bonding agent in primary molars with a 12-month follow-up. A total of 40 patients aged 5-9 years with at least two dentin caries (D1 Level) in primary molars were included in the study. The study involved a split-mouth design in which Ultradent PQ1 Bond and Ultradent Peak Universal Bond were used as the bonding agents and Tetric N Ceram Bulk Fill composite was used as the restorative material for the restoration of primary molars with class II cavity. The evaluation of clinical success was performed by a calibrated observer according to the FDI criteria at months 3, 6, 9, and 12 after restoration.

ELIGIBILITY:
Inclusion Criteria:

(1) age between 5-9 years; (2) no systemic health problems (3) presence of at least one interproximal carious lesion not exceeding half of the dentin structure (D1 level) in the right and left sides of the mouth; (4) cooperation without issues (scoring 3 or 4 on the Frankl scale); and (5) patient and parent's willingness to attend follow-up appointments throughout the study.

Exclusion Criteria:

* (1) the presence of pulp vitality with no clinical and/or radiological signs requiring endodontic treatment, (2) no previous treatment on the selected teeth, (3) Radiographically, the caries should not extend to one-third of the pulp, indicating only the need for a Class II restoration, (4) the presence of adjacent teeth mesial and distal to the selected tooth and an opposing tooth in the oral cavity, (5) the absence of physiological or pathological root resorption.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | The treatments will be assessed using the same method over a 12-month period with 3-month intervals.
  Following the completion of the restorations, a proficient observer, unaware of the utilized material, will assess the respective tooth based on the World Dental Federation (FDI) criteria (reference). This evaluation will be conducted using a mirror and probe under illumination, with teeth being dried using air/water spray. The assigned scores will categorize the restorations as successful (Score 1), exhibiting minor defects (Score 2), showing acceptable defects (Score 3), needing repair (Score 4), or necessitating replacement (Score 5).

IPD SHARING:
Plan to Share IPD: No
there are no plans to make individual participant data (IPD) available to other researchers.